CLINICAL TRIAL: NCT03828123
Title: A Prospective, Non-randomized, Open Label Study to Assess the Safety and the Efficacy of Autologous Multipotent Mesenchymal Stromal Cells in the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Autologous Multipotent Mesenchymal Stromal Cells in the Treatment of Amyotrophic Lateral Sclerosis
Acronym: AMSC-ALS-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bioinova, s.r.o. (Industry)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMSC-ALS-001
Record Dates: First submitted 2017-07-20; First posted 2019-02-04 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Multipotent MSC (Experimental): Patients with intrathecal administration of Suspension of human autologous MSC 3P in 1.5 ml
  Interventions: Biological: Suspension of human autologous MSC 3P in 1.5 ml

INTERVENTIONS:
Biological: Suspension of human autologous MSC 3P in 1.5 ml — Intrathecal application of Autologous Multipotent Mesenchymal Stromal Cells 3P suspension

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a progressive neurodegenerative disease that targets motor neurons. Prognosis is invariably fatal within 3-5 years since manifestation of the disease. Despite improved understanding of the mechanisms underlying ALS, the treatment remains essentially only supportive and focused on symptoms relief. Over the past few years, stem cell research has expanded greatly as a tool for developing new therapies to treat incurable diseases. Stem cell therapy has been shown as promising in several animal ALS models and human clinical trials.

DETAILED DESCRIPTION:
Subjects will be assigned to autologous mesenchymal stromal cell (AMSC) treatment according to inclusion and exclusion criteria (see below) screened four times prior to administration. Then the subjects will be observed for three consecutive yearsAfter a half year of screening period, the autologous multipotent mesenchymal stromal cells from bone marrow will be isolated. The cells will be cultivated for 3 passages (3 - 4 weeks) in order to get sufficient amount for therapy, cell suspension for intrathecal application will be prepared and introduced intrathecally through lumbar puncture. Subsequently, all the subjects will be observed at the range of standard medical care used at these types of interventions.

ELIGIBILITY:
Inclusion Criteria:

1. established diagnosis of definite ALS according to El Escorial criteria
2. riluzole naive or stable dose for at least 2 months,
3. life expectancy more than 2 years
4. patients able to provide written informed consent.

Exclusion Criteria:

1. FVC less than 70%
2. in case of primary bulbar paralysis less than 15 points on Norris bulbar scale,
3. less than 15 points on Norris spinal scale,
4. pregnancy, breastfeeding
5. coagulopathy,
6. skin infection at the site of bone marrow aspiration or application of the cell product,
7. gastrostomy,
8. any significant medical condition that would compromise the safety of the patient (e.g. recent myocardial infarction, congestive heart failure, renal failure, liver failure, cancer, systemic infection, recurrent thromboembolic disease .....),
9. alcohol or drug abuse
10. cancer.
11. women of childbearing potential not using effective contraception (established oral contraception, intrauterine device, ligation of the uterine tube) including proven contraceptive measures taken by their sexual partners
12. fertile men not using proven contraceptive measures including effective contraception of their partner (established oral contraception, intrauterine device, ligation of the uterine tube)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Safety: Complications related to the medicinal product application - new neurological deficit and occurrence of other adverse events | 1 year
  Complications at the site of intrathecal infusion of the medicinal product and no new neurological deficit (meningism, paraplegia, urinary incontinence) not attributed to the natural progression of the ALS disease will be recorded at Visits I, III, IV, V, VI, and IX. Occurrence of other potential adverse events, including headache, respiratory failure, leukocytosis, cervical spine stenosis, cystitis and hyperhydrosis will be evaluated on the severity scale (1=mild, 2=moderate, 3=severe).
  Brain and spinal cord MRI will be performed at Visits I and IX to exclude treatment-related tumor formation, pathological contrast enhancement or other structural pathology.

SECONDARY OUTCOMES:
Efficacy: Inhibition of the disease progression - ALS functional rating scale | 18 months
  Inhibition of the disease progression will be recorded by ALS functional rating scale (ALSFRS) at Visits I, III, and VI through X.
  Measures (all 4-0):
  1. speech
  2. salivation
  3. swallowing
  4. handwriting
  5. cutting food and handling utensils (with or without gastrostomy)
  6. dressing and hygiene
  7. turning in bed and adjusting bed clothes
  8. walking
  9. climbing stairs
  10. breathing
  ALSFRS = SUM (points for all 10 measures)
  Interpretation:
  minimum score: 0 maximum score: 40 The higher the score the more function is retained.
Efficacy: Inhibition of the disease progression - Norris scale | 18 months
  Inhibition of the disease progression will be recorded by Norris scale at Visits I, III, and VI through X.
  Norris scal has has 22 items examining bulbar, respiratory, trunk, arm, leg, and general domains involving reflexes, fasciculation, and muscle atrophy. The scale also measures emotional lability, fatigability and leg rigidity. The Norris scale has a linear decline during the course of ALS.
Efficacy: Inhibition of the disease progression - Forced vital capacity (FVC) | 18 months
  FVC (%) will be measured at Visits I, and VI through X.

REFERENCES:
- [Result] Sykova E, Rychmach P, Drahoradova I, Konradova S, Ruzickova K, Vorisek I, Forostyak S, Homola A, Bojar M. Transplantation of Mesenchymal Stromal Cells in Patients With Amyotrophic Lateral Sclerosis: Results of Phase I/IIa Clinical Trial. Cell Transplant. 2017 Apr 13;26(4):647-658. doi: 10.3727/096368916X693716. Epub 2016 Nov 7. PMID 27938483